CLINICAL TRIAL: NCT00533780
Title: Effect of Healing Touch on the Experience of Women Undergoing Treatment for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Avon Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRSADJ0003; 95738 (Other: Stanford University Alternate IRB Number); 14064 (Other: Stanford IRB)
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI high resolution 3D diffusion (Experimental): Total duration is about 8 minutes.
  Interventions: Procedure: Healing Touch

INTERVENTIONS:
Procedure: Healing Touch — A gentle, non-invasive form of energy-balancing work that promotes relaxation and can help manage the side effects of chemotherapy.

SUMMARY:
To learn what effect, if any, Healing Touch (a gentle, non-invasive form of energy work that promotes relaxation and can help manage the side effects of chemotherapy and radiation), has on physical symptoms, mood, and qualify of life for women undergoing treatment for breast cancer.

ELIGIBILITY:
Inclusion Criteria:- Patients undergoing treatment for breast cancer.

* Age 18 or over.
* Participants in Healing Partners Program. Exclusion Criteria:- Patients not under the care of a physician.
* Patients not able to come to regular healing touch sessions.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn M Westphal, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healing Touch: Healing Touch : A gentle, non-invasive form of energy-balancing work that promotes relaxation and can help manage the side effects of chemotherapy.
Period: Overall Study
Arm/Group | Healing Touch
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healing Touch
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: FACT-B Quality of Life Score
Description: Final scores (FACT-B-Total) of all subscales range from 0 to 148, where 148 represents the most favorable score and accordingly a highest QoL.
Time Frame: month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healing Touch
Number analyzed (Participants) | 51
score on a scale | 91.9 (17.6)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Healing Touch
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes